CLINICAL TRIAL: NCT06975384
Title: The Associations of Sleep Disturbance With Therapy Efficacy and Prognosis of Lung Cancer, Including Non-small-cell Lung Cancer and Small-cell Lung Cancer With Early and Advanced Staging
Brief Title: The Associations of Sleep Disturbance With Therapy Efficacy and Prognosis of Lung Cancer
Acronym: Nezha
Status: Recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Fang Wu, Professor, Second Xiangya Hospital of Central South University
Other Study IDs: LYF20240270
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer; Sleep Disturbance; Immune Checkpoint Inhibitors; Cancer, Treatment-Related
Keywords: Lung Cancer; Immune Checkpoint Inhibitors; Sleep Disturbance; Circadian Rhythm; Cancer Progression; Prognosis; Biomarker
MeSH Terms: conditions — Lung Neoplasms; Parasomnias; Neoplasms, Second Primary; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — baseline tumor tissue, serial blood and stool samples (baseline and treatment follow-up time points).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Advanced NSCLC patients receiving first-line ICIs: For stage IIIB-IV patients with NSCLC who have received immune checkpoint inhibitors as first-line therapy.
  Interventions: Other: Exposure: sleep disturbance status
- Limited-stage and extensive-stage SCLC patients receiving first-line ICIs: For limited-stage and extensive-stage SCLC patients who have received immune checkpoint inhibitors as first-line therapy.
  Interventions: Other: Exposure: sleep disturbance status
- NSCLC patients receiving neoadjuvant therapy of ICIs: For stage IB-IIIB patients with non-small cell lung cancer who have received neoadjuvant therapy of immune checkpoint inhibitors.
  Interventions: Other: Exposure: sleep disturbance status
- Early stage NSCLC patients receiving radical resection: For early-stage patients with non-small cell lung cancer who have received radical resection.
  Interventions: Other: Exposure: sleep disturbance status
- Advanced NSCLC patients receiving first-line targeted therapy: For stage IIIB-IV patients with NSCLC who have received targeted agents as first-line therapy.
  Interventions: Other: Exposure: sleep disturbance status

INTERVENTIONS:
Other: Exposure: sleep disturbance status — The assessment of sleep disturbance was conducted using Pittsburgh Sleep Quality Index (PSQI) and Insomnia Severity Index (ISI). Patients with a PSQI score > 5 or an ISI score > 7 were categorized as sleep disturbance patients.
  The assessment of chronotype was conducted using reduced Morningness-Eveningness Questionnaire (rMEQ). Patients with an rMEQ score 18-25 were categorized as the morning type, those with an rMEQ score 12-17 as the intermediate type, and those with an rMEQ score 4-11 as the evening type.

SUMMARY:
This is the prospective, observational cohort study (Nezha) to explore the associations of sleep disturbance with progression, efficacy of immune checkpoint inhibitors (ICIs) and prognosis of Lung Cancer. The participants including the patients diagnosed with advanced non-small-cell lung cancer (NSCLC) who received either first-line therapy (ICIs or targeted agents) or neoadjuvant therapy with ICIs; patients diagnosed with advanced small-cell lung cancer (SCLC) receiving the first-line therapy ICIs; patients diagnosed with early non-small-cell lung cancer (NSCLC) receiving surgery.

DETAILED DESCRIPTION:
This is the prospective, observational cohort study (Nezha) to explore the associations of sleep disturbance with progression, efficacy of ICIs and prognosis of Lung Cancer. This study will have 5 cohorts

* Cohort 1: A prospective, observational cohort study to explore the association between sleep disturbance and the efficacy of first-line treatment of ICIs in advanced NSCLC.
* Cohort 2: A prospective, observational cohort study to explore the association between sleep disturbance and the efficacy of first-line treatment of limited-stage and extensive-stage SCLC.
* Cohort 3: A prospective, observational cohort study to explore the association between sleep disturbance and the efficacy of neoadjuvant therapy of ICIs in resectable NSCLC.
* Cohort 4: A prospective, observational cohort study to explore the association of sleep disturbance with postoperative recurrence and prognosis in early-stage NSCLC receiving radical surgery.
* Cohort 5: A prospective observational cohort study to explore the association between sleep disturbance and the efficacy of first-line treatment of targeted therapy in advanced NSCLC.

ELIGIBILITY:
Cohort 1:

Inclusion Criteria:

1. Age ≥ 18 years old;
2. Histologically confirmed diagnosis of NSCLC;
3. Unresectable locally advanced, metastatic, or recurrent stage ⅢB-Ⅳ based on AJCC TNM staging 8th edition;
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1;
5. Treatment naïve;
6. Presence of at least one measurable lesion according to the Response Evaluation Criteria in Advanced Solid Tumors version 1.1 (RECIST v1.1);
7. Receiving PD-1/PD-L1 inhibitors monotherapy or combination with chemotherapy;
8. Informed consent to participate in the study;

Exclusion Criteria:

1. Epidermal growth factor receptor (EGFR)-sensitizing mutation and/or anaplastic lymphoma kinase (ALK) fusion and/or ROS proto-oncogene 1 (ROS1) fusion-positive;
2. Presence of other malignant tumors or malignant diseases within 3 years;
3. Concurrent acute or chronic psychiatric disorders;
4. Patients receiving sleep medication;
5. Prior participation in other clinical drug trials;
6. Symptomatic brain metastasis;
7. Inability to complete scale assessments.

Cohort 2:

Inclusion Criteria:

1. Age ≥ 18 years old;
2. Histologically confirmed diagnosis of SCLC；
3. Unresectable locally advanced, metastatic, or recurrent stage Ⅲ-Ⅳ based on AJCC TNM staging 8th edition;
4. ECOG PS of 0-1;
5. Treatment naïve;
6. Presence of at least one measurable lesion according to the RECIST v1.1 ;
7. Receiving PD-1/PD-L1 inhibitors monotherapy or combination with chemotherapy;
8. Informed consent to participate in the study;

Exclusion Criteria:

1. Presence of other malignant tumors or malignant diseases within 3 years;
2. Concurrent acute or chronic psychiatric disorders;
3. Patients receiving sleep medication;
4. Prior participation in other clinical drug trials;
5. Symptomatic brain metastasis;
6. Inability to complete scale assessments.

Cohort 3:

Inclusion Criteria:

1. Age ≥18 years old;
2. Pathologically diagnosed as NSCLC;
3. Resectable clinical stage IB-IIIB based on AJCC TNM staging 8th edition;
4. At least one measurable lesion can be evaluated according to the RECIST v1.1;
5. Treatment naïve;
6. Receiving PD-1/PD-L1 inhibitors monotherapy or combination with chemotherapy as neoadjuvant therapy;
7. Cardiopulmonary function can withstand surgery;
8. Informed consent to participate in the study.

Exclusion Criteria:

1. EGFR-sensitizing mutation and/or ALK fusion and/or ROS1 fusion-positive;
2. Presence of other malignant tumors or malignant diseases within 3 years;
3. Concurrent acute or chronic psychiatric disorders;
4. Patients receiving sleep medication;
5. Prior participation in other clinical drug trials;
6. Symptomatic brain metastasis;
7. Inability to complete scale assessments.

Cohort 4:

Inclusion Criteria:

1. Age ≥ 18 years old;
2. Pathologically diagnosed as NSCLC;
3. Pathologically stage confirmed as early stage of IA-IIIA;
4. Available for tumor tissue samples;
5. Treatment naïve;
6. Receiving radical surgery;
7. Informed consent to participate in the study;

Exclusion Criteria:

1. Presence of other malignant tumors or malignant diseases within 3 years;
2. Concurrent acute or chronic psychiatric disorders;
3. Patients receiving sleep medication;
4. Prior participation in other clinical drug trials;
5. Inability to complete scale assessments.

Cohort 5:

Inclusion Criteria:

1. Age ≥ 18 years old;
2. Histologically confirmed diagnosis of NSCLC;
3. Unresectable locally advanced, metastatic, or recurrent stage ⅢB-Ⅳ based on AJCC TNM staging 8th edition;
4. ECOG PS of 0-1;
5. Treatment naive;
6. Presence of at least one measurable lesion according to the RECIST v1.1;
7. Receiving targeted therapy or combination with chemotherapy;
8. Informed consent to participate in the study;
9. Driver gene-positive.

Exclusion Criteria:

1. Presence of other malignant tumors or malignant diseases within 3 years;
2. Concurrent acute or chronic psychiatric disorders;
3. Patients receiving sleep medication;
4. Prior participation in other clinical drug trials;
5. Symptomatic brain metastasis;
6. Inability to complete scale assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants including the patients diagnosed with advanced non-small-cell lung cancer (NSCLC) who received either first-line therapy (ICIs or targeted agents) or neoadjuvant therapy with ICIs; patients diagnosed with advanced small-cell lung cancer (SCLC) receiving the first-line therapy ICIs; patients diagnosed with early non-small-cell lung cancer (NSCLC) receiving surgery.
Sampling Method: Probability Sample
Enrollment: 1270 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Cohort 1 & 5: Progression-free survival (PFS) | 3 years
  Time from the beginning of first-line immunotherapy or targeted therapy to the first progression (PD).
Cohort 2: Overall survival (OS) | 5 years
  Duration from the beginning of first-line immunotherapy until death due to any cause. Subjects who are still alive at the end of the study observation period will be censored at the time of last known vital status.
Cohort 3: Event-free survival (EFS) | 3 years
  Time from the start of initial treatment of immunotherapy to the occurrence of any event, including disease progression, discontinuation of treatment for any reason, or death.
Cohort 4: Disease-free survival (DFS) | 5 years
  Duration between the date after surgery to the date of any recurrence or death firstly.

SECONDARY OUTCOMES:
Cohort 2: Progression-free survival (PFS) | 3 years
  Time from the beginning of first-line immunotherapy to the first progression (PD).
Cohort 1 & 3 & 4 & 5: Overall survival (OS) | 5 years
  Overall Survival (OS) is defined as the duration from the start of initial treatment (systemic treatment or radical therapy) until death from any cause. Subjects who are still alive at the end of the study observation period will be censored at the time of last known vital status.
Quality of life (QoL) | 5 years
  Quality of life (QoL) is assessed longitude by EORTC QLQ-C30 (version.3). The EORTC QLQ-C30 is composed of 9 multi-item scales: 5 functioning scales (physical, role, cognitive, emotional, and social), a global QOL scale, and 3 symptom scales (fatigue, pain, and nausea/vomiting). All scales and single items are linearly transformed to an 0-100 scale. A higher score represents a better level of functioning.
Cohort 1 & 2 & 5: Objective Response Rate (ORR) | 2 years
  The proportion of patients with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Cohort 3: Pathologic complete response (pCR) rate | 3 years
  pCR is no viable tumor cells in tumor bed and lymph nodes. The pCR rate is the proportion of patients with a pathologic complete response.
Cohort 3: Major pathologic response (MPR) | 3 years
  MPR refers to the percentage of surviving tumor cells in the tumor bed after neoadjuvant therapy ≤10%, regardless of whether there are surviving tumor cells in the lymph nodes.

OTHER OUTCOMES:
Gut microbiota signature | 5 years
  The baseline fetal is collected and assessed by 16S rRNA sequencing to explore the association between gut microbiota, states of sleep disturbance and efficacy and prognosis.
Tumor microenvironment signature | 5 years
  The baseline paraffin-embedded tissue is collected and assessed by multiplex immunohistochemistry, single-cell sequencing, and spatial transcriptome sequencing to explore the association between tumor microenvironment signature, states of sleep disturbance and efficacy and prognosis.
Peripheral blood biomarker and immune cells signature | 5 years
  The baseline peripheral venous blood is collected. Sleep-related biomarkers (including melatonin, epinephrine, norepinephrine, cortisol, serotonin, dopamine, and endorphins) are measured. The peripheral immune cells signature is assessed by flow cytometry, including T lymphocytes, B lymphocytes, NK lymphocytes, macrophagocyte, and dendritic cells (DCs). And explore the associations between peripheral blood biomarkers, immune cells signature, states of sleep disturbance and efficacy and prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, The Second Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No